CLINICAL TRIAL: NCT00244855
Title: Rituximab and Dexamethasone in CD20 Positive Low Grade and Follicular Non-Hodgkin's Lymphoma
Brief Title: Rituximab and Dexamethasone in Treating Patients With Low-Grade Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Maloney, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSOC 2002; NCI-2011-00576 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Marginal Zone Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Marginal Zone Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Waldenstrom Macroglobulinemia | interventions — Rituximab; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No previous treatment (Other): Patients received no previous treatment. Patients enrolled in the trial received dexamethasone IV and rituximab IV once weekly. Treatment continues for 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: pharmacological study; Biological: rituximab; Drug: dexamethasone; Other: laboratory biomarker analysis
- Previous treatment (Other): Patients received previous treatment. Patients enrolled in the trial received dexamethasone IV and rituximab IV once weekly. Treatment continues for 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: pharmacological study; Biological: rituximab; Drug: dexamethasone; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: dexamethasone — Given IV
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well giving rituximab and dexamethasone together works in treating patients with low-grade non-Hodgkin lymphoma (NHL). Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with dexamethasone may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate clinical response rate (RR) at 3 and 6 months. II. To estimate Grade 2-4 -infusion-related toxicity.

SECONDARY OBJECTIVES:

I. To evaluate laboratory parameters and correlate with clinical response including: antibody dependent cell mediated cytotoxicity and effector cell phenotype analysis at baseline, 4 weeks and three months.

II. To evaluate laboratory parameters and correlate with clinical response including: soluble cluster of differentiation (CD)20 fragments or CD20-containing membrane fragments at baseline, 4 weeks, and 3 months.

III. To evaluate laboratory parameters and correlate with clinical response including: phenotype analysis of CD16 and CD32 on natural killer (NK) cells.

IV. To evaluate laboratory parameters and correlate with clinical response including: rituximab pharmacokinetic studies at baseline, 4 weeks and 3 months.

OUTLINE:

Patients receive dexamethasone intravenously (IV) and rituximab IV once weekly. Treatment continues for 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven CD20+ low grade B cell lymphoma including follicular, marginal zone, monocytoid B cell, and lymphoplasmacytoid lymphoma; patients may be previously untreated or in relapse
* Patients must have measurable disease with clearly defined margins assessed by physical exam with direct measurement (for cutaneous B-cell lymphomas), computed tomography (CT) or magnetic resonance imaging (MRI), defined as >= 20 mm with conventional CT or MRI or >= 10 mm using spiral CT scan
* Absolute neutrophil count >= 1000/mm^3
* Hemoglobin > 7 g/dl
* Platelets >= 100,000/mm^3
* Serum creatinine =< 2.5 mg/dl
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2x the upper limit of normal (ULN)
* Karnofsky performance score >= 70 %
* Patient has signed an Institutional Review Board (IRB) approved informed consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Patient has received rituximab therapy within 6 months of entry into protocol
* Patient has received systemic steroid therapy within one month of entry into protocol
* Patient has Intermediate or High Grade NHL, mantle cell lymphoma, chronic lymphocytic leukemia, or small lymphocytic lymphoma
* Patient is pregnant or lactating
* Patient is unwilling or unable to practice contraception during treatment and for one year thereafter
* Patient has active central nervous system (CNS) disease
* Patient has human immunodeficiency virus (HIV) disease
* Patient has an active infection requiring antimicrobial therapy
* Patient has significant heart disease, New York Heart Classification III or IV heart disease (III: Marked limitation of physical activity; comfortable at rest, but less than ordinary activity causes fatigue, or dyspnea; IV: Unable to carry on any physical activity without symptoms; symptoms are present even at rest; if any physical activity is undertaken, symptoms are increased)
* Patient requires supplemental oxygen
* Patient has a concomitant malignancy or previous malignancy within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, or in situ cervical or in situ breast cancer
* Patients with active hepatitis B virus (HBV) infection or hepatitis, or with hepatitis C positive serology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2011-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Previous Treatment | Previous Treatment
Started | 7 | 25
Completed | 7 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Previous Treatment | No Previous Treatment | Total
Number analyzed (Participants) | 7 | 25 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 14 | 17
  >=65 years | 4 | 11 | 15
Age, Continuous [Median (Full Range); unit: years] | 67 [42 to 79] | 64 [38 to 85] | 64 [38 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 17 | 21
  Male | 3 | 8 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 6 | 23 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 25 | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Survival without measurable progression of lymphoma estimated according to the Kaplan-Meier method
Time Frame: At 3 and 6 months after enrollment
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier estimated % of patients
Arm/Group | Previous Treatment | No Previous Treatment
Number analyzed (Participants) | 7 | 25
Kaplan-Meier estimated % of patients
  At 3 months after enrollment | 92 [81 to 100] | 71 [45 to 100]
  At 6 months after enrollment | 83 [70 to 100] | 71 [45 to 100]

2. Secondary Outcome: Survival
Description: Percentage of patients remaining alive estimated according to the Kaplan-Meier method
Time Frame: At 6 months, 12 months and 24 months after enrollment
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier estimated % of patients
Arm/Group | No Previous Treatment | Previous Treatment
Number analyzed (Participants) | 7 | 25
Kaplan-Meier estimated % of patients
  At 6 months | 96 [88 to 100] | 100 [100 to 100]
  At 12 months | 96 [88 to 100] | 100 [100 to 100]
  At 24 months | 91 [80 to 100] | 67 [38 to 100]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Previous Treatment | No Previous Treatment
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/25
Other Adverse Events (participants affected / at risk) | 5/7 | 16/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Previous Treatment (N=7) | No Previous Treatment (N=25)
Vasovagal episode (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Cardiac disorders) | 1 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 1
Lymphopenia (Immune system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0
Urticaria (Immune system disorders) | 1 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Penile infection (Infections and infestations) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 3
Confusion (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 1
Pain (General disorders) | 1 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Sweating (General disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperglycemia (Endocrine disorders) | 0 | 1
Hypoglycemia (Endocrine disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes